CLINICAL TRIAL: NCT03000517
Title: Pharmacokinetics of Levofloxacin in MDR-TB Patients
Brief Title: PK of Levofloxacin in MDR-TB Patients
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jan-Willem C Alffenaar, PhD PharmD Clinical Pharmacologist, University Medical Center Groningen
Other Study IDs: LFX/V0.1
Record Dates: First submitted 2016-09-01; First posted 2016-12-22 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Multi-drug Resistant Tuberculosis
Keywords: levofloxacin; multi-drug resistant TB; pharmacokinetics
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and saliva samples of MDR-TB patients on 0 hr premedication and 1,2,4,8 hrs post mediation.
Oversight: Data Monitoring Committee: No

SUMMARY:
The emergence and spread of multi-drug resistant and extensively-drug resistant strains of Mycobacterium tuberculosis (MDR/XDR-TB) have posed a great threat to global TB control and elimination, limiting treatment success rate at worrisome 50% for MDR-TB. Among various factors contributing to the development of drug resistance, low drug exposure is well recognized. To overcome this, either new drugs have to be developed or the dose of currently used therapy be optimized, or both. Fluoroquinolones (levofloxacin and moxifloxacin) and aminoglycosides are important drugs in the MDR-TB treatment regimen. Development of acquired drug resistance to these drugs could complicate and narrow down the available options, and further exacerbate to pre-XDR and XDR-TB.

Objective:

The main objective of this prospective clinical study is to understand the pharmacokinetics of levofloxacin in MDR-TB patients, receiving standard dosage (750-1250mg) based on the body weight and correlate drug exposure, with treatment outcomes.

Study design:

A prospective pharmacokinetic study

Study population: 20 MDR-TB patients

Intervention: Patients receive once daily oral dosing of levofloxacin (750-1250mg) based on the body weight, under MDR-TB treatment regimen of Nepal.

Main study parameters/end points:

The pharmacokinetic parameters(Vd, CL, AUC etc.) of levofloxacin are the primary end points of the study. The Cmax/MIC and AUC0-24h/MIC ratios are the best predictive parameters for efficacy of levofloxacin treatment and will be estimated. Pharmacokinetics will be evaluated in plasma and in oral fluid

ELIGIBILITY:
Inclusion Criteria:

* Patient with TB, with Mycobacterium tuberculosis by culture/ Gene Xpert
* Patient is 18 years or older with newly diagnosed or previously treated MDR-TB
* Patient with sputum smear positive for acid-fast bacilli or sputum smear negative but Gene Xpert (MTB/RIF) positive, and resistant to both isoniazid and rifampicin
* Patients with MDR-TB receiving levofloxacin as a part of MDR-TB regimen

Exclusion Criteria:

* Patient with neurologic or severe extra-pulmonary manifestations of tuberculosis
* Pregnant women or breast feeding mothers with MDR-TB
* Patients with diminished renal functions or on medications for the treatment of renal disorders
* Body weight <35 kg
* Patients treated with aluminium- and magnesium containing antacids and ferrous sulphates, cimetidine and probenecid, theophylline, warfarin, zidovudine, digoxin or cyclosporine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with previously treated or newly diagnosed MDR-TB who are at the end of first month(15-30th day) and second month (45-60th day) of their treatment.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
AUC | Period I (15-30) day and Period II (45-60) day
  The main objective of this prospective clinical trial is to evaluate the levofloxacin exposures (AUC) of a standard dose (750-1250mg) in plasma and saliva of MDR-TB patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Willem Alffenaar, Principal Investigator — University Medical Center Groningen, University of Groningen
Locations (1):
- German Nepal Tuberculosis Project Clinic (GENETUP), Kalimati, Kathmandu, Nepal

REFERENCES:
- [Derived] Ghimire S, Maharjan B, Jongedijk EM, Kosterink JGW, Ghimire GR, Touw DJ, van der Werf TS, Shrestha B, Alffenaar JC. Evaluation of Saliva as a Potential Alternative Sampling Matrix for Therapeutic Drug Monitoring of Levofloxacin in Patients with Multidrug-Resistant Tuberculosis. Antimicrob Agents Chemother. 2019 Apr 25;63(5):e02379-18. doi: 10.1128/AAC.02379-18. Print 2019 May. PMID 30782999